CLINICAL TRIAL: NCT03630809
Title: Immune Response Surveillance and Potential Booster Vaccines for Patients Who Have Received HER2-pulsed DC1 Vaccine
Brief Title: Immune Response and Potential Booster for Patients Who Have Received HER2-pulsed DC1
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Quality of the data originating from prior versions of the protocol has been affected by protocol deviations triggered by the COVID-19 pandemics
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-19650
Record Dates: First submitted 2018-08-10; First posted 2018-08-15 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Breast Cancer; HER2-positive Breast Cancer; HER-2 Gene Amplification; HER2 Positive Breast Carcinoma; HER-2 Protein Overexpression; Breast Cancer, Male; Breast Cancer Female
Keywords: nonmetastatic; classic HER2; Nonmetastatic classic HER2
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Previously enrolled in study or have been previously treated with DC1 Vaccines - Arm A (Active Comparator): Participants currently enrolled into arm A will offered randomization into arms C or D. If study participants decline randomization or are ineligible, they will complete study follow up visits as stated in the schedule of events per Arm A.
  Interventions: Biological: HER2 DC1 Vaccine
- Participants receiving first 3 boosters at 3 month intervals - Arm B (Active Comparator): A history and physical exam will be taken at 3-month intervals. Any changes in history or physical condition will be documented. Patient currently enrolled into arm B will offered randomization into arms C or D once finished with arm B. If patients decline randomization or are ineligible, they will complete study follow up visits as stated in the schedule of events per Arm B.
  Interventions: Biological: HER2 DC1 Vaccine
- Participants receiving 3 booster vaccines at 3-month intervals (+/- 30 days window) - Arm C (Experimental): A history and physical exam will be taken at 3-month intervals. Any changes in history or physical condition will be documented
  Interventions: Biological: HER2 DC1 Vaccine
- Participants receiving 6 booster vaccines at 3-month intervals (+/- 30 days window) - Arm D (Experimental): A history and physical exam will be taken at 3-month intervals. Any changes in history or physical condition will be documented.
  Interventions: Biological: HER2 DC1 Vaccine

INTERVENTIONS:
Biological: HER2 DC1 Vaccine — Ultrasound (US) guided intranodal delivered vaccines will be administered at each participating site by a radiologist experienced in ultrasound guided procedures along with the principal investigator or his/her designee. Each dose will consist of between 1.0-2.0 x 10^7 cells and will be injected into 1 right and 1 left normal groin lymph nodes.
  Other Names: Vaccine

SUMMARY:
The purpose of this study is to learn more about how to treat patients with a diagnosis of diagnosis of Human Epidermal Growth Factor Receptor 2/neu (HER-2/neu) positive breast cancer in the past, who were previously treated with HER-2/neu-directed dendritic cells (DC) vaccines.

There is evidence that the use of anti-HER2 dendritic cell (DC) study vaccines could improve response to breast cancer therapy and be an important step in the prevention of recurrence.

This study will use a Dendritic Cell Type 1 (DC1) vaccine which is a HER2-sensitized dendritic cell (DC) study vaccine. Dendritic cells are immune cells that can tell the participant's immune system to fight infection. This study vaccine will be made from the participant's blood cells collected from a procedure called leukapheresis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of nonmetastatic or metastatic breast cancer in complete clinicla response classic HER2pos (ie, IHC 3+ or FISHpos) breast cancer (BC) who have previously been vaccinated with DC1 HER2-pulsed vaccines on any of several prior clinical trials for ductal carcinoma in situ (DCIS) or inflammatory breast cancer (IBC) are eligible; however, we also allowed HER2 2+ patients in many of these prior trials and they will also be allowed to participate in this trial. Note: HER2pos BC is defined by tumor tissue HER2 overexpression and or tumor HER2 amplification. The lack of HER2 overexpression by IHC is defined as 0 or 1+ whereas overexpression is defined as 3+. In the event of equivocal IHC, 2+, the tumor must be gene-amplified by fluorescent in situ hybridization (FISH) performed upon the primary tumor or metastatic lesion (ratio > 2 and HER2 copy number > 4 define HER2negdisease).
* Patients with nonmetastatic HER posBC must have completed all standard-of-care treatment for nonmetastatic BC (e.g., surgery, chemotherapy, radiation therapy, and HER2-targeted therapy). Note: antiestrogen therapy is permitted while on trial. Note: antiestrogen therapy is permitted while on trial.
* Patients with diagnosis of metastatic HER2 pos breast cancer must have complete tumor response to current treatment per RECIST 1.1 and completed all standard-of-care chemotherapy. Note: maintenance treatment with approved HER2-targeted agents and/or antiestrogen therapy is permitted while on trial.
* Age ≥ 18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
* Participants must have normal organ and marrow function within 2 weeks of registration.
* For both male and female patients, effective methods of contraception must be used throughout the study and for 3 months following the last dose.
* Must have the ability to understand and the willingness to sign a written informed consent prior to registration on study.

Exclusion Criteria:

* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, congenital prolonged QT syndrome, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Uncontrolled congenital or acquired immune deficiency that is requiring treatment that would interfere with study treatment will not be allowed on study. Topical, ocular, intra-articular, intranasal, inhalational corticosteroids (with minimal systemic absorption) are allowed. Patients who have received systemic corticosteroids ≤ 30 days prior to starting study drug will be excluded.
* No other prior malignancy is allowed except for the following:

  * Adequately treated basal cell or squamous cell skin cancer
  * In situ cervical cancer
  * Any other cancer from which the patient has been disease free for at least 3 years.
* Pregnant or breast feeding.
* Known to be HIV positive.
* Known current or a history of hepatitis B or C virus, including chronic and dormant states, unless disease has been treated and confirmed cleared.
* Major surgery within 4 weeks of initiation of study drug.
* Have not recovered to ≤ Grade 1 or tolerable Grade 2 adverse events (AEs) due to agents administered ≥ 28 days earlier, as documented by the treating investigator.
* Currently enrolled in any other clinical protocol or investigational trial that involves administration of experimental therapy and/or therapeutic devices, or investigational drug. Note: patients enrolled on another HER2 vaccine trial but not receiving active therapy can enroll in this study.
* Not able to comply with the treatment schedule and study procedures for any reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2022-04-11 (Actual); Study Completion 2022-04-11 (Actual)

PRIMARY OUTCOMES:
HER2 DC1 Vaccine Regimen | Up to 16 months
  Investigators will assess the feasibility of participants receiving the six-booster regimen if 11/15 randomized to Arm D complete all 6 booster injections.

SECONDARY OUTCOMES:
HER2 Immunity with 3 Booster Regimen at 18 months | At 18 months after first dose
  To compare the overall average effects of two different vaccine regimens on anti-HER2 CD4 immunity (ELISPOT) at 18 months from month 1 injection. treatment among women with breast cancer previously treated with HER2 vaccines. Two regimens consist of 3 versus 6 booster HER2 vaccine injections administered every 3 months
HER2 Immunity with 6 Booster Regimen at 18 months | At 18 months after first dose
  To compare the overall average effects of two different vaccine regimens on anti-HER2 CD4 immunity (ELISPOT) at 18 months from month 1 injection. treatment among women with breast cancer previously treated with HER2 vaccines. Two regimens consist of 3 versus 6 booster HER2 vaccine injections administered every 3 months
HER2 Immunity with 3 Booster Regimen at 10 months | At 10 months after first dose
  To compare the overall average effects of two different vaccine regimens on anti-HER2 CD4 immunity (ELISPOT) at month 10 from first vaccine treatment
HER2 Immunity with 6 Booster Regimen at 10 months | At 10 months after first dose
  To compare the overall average effects of two different vaccine regimens on anti-HER2 CD4 immunity (ELISPOT) at month 10 from first vaccine treatment
Rate of Treatment Emergent Adverse Events of 3 Dose Regimen | Up to 5 years
  Serious adverse events will be recorded for 100 days after study treatment. Adverse events will follow National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Rate of Treatment Emergent Adverse Events of 6 Dose Regimen | Up to 5 years
  Serious adverse events will be recorded for 100 days after study treatment. Adverse events will follow National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Overall Survival | Up to 5 Years
  OS will be measured using the Kaplan-Meier method
Disease Free Survival | Up to 5 Years
  DFS will be measured using the Kaplan-Meier method
Progression Free Survival | Up to 5 Years
  PFS will be measured using the Kaplan-Meier method

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Costa, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States